CLINICAL TRIAL: NCT01443468
Title: Clinical, Epidemiologic, and Genetic Studies of Li-Fraumeni Syndrome
Brief Title: Clinical and Genetic Studies of Li-Fraumeni Syndrome
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110255; 11-C-0255
Record Dates: First submitted 2011-09-28; First posted 2011-09-29 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-12-05

CONDITIONS: Li-Fraumeni Syndrome; Neoplasms; Tp53 Mutations
Keywords: Tp53; Cancer; Hereditary; Genetic Testing; Screening
MeSH Terms: conditions — Li-Fraumeni Syndrome; Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 1: Patients within a family with a known TP53 mutation who are positive for that mutation.
- 2: Patients within a family with a known TP53 mutation who are negative for that mutation.
- 3: Unaffected family members.
- 4: Patients who meet clinical LFS criteria but haven't had TP53 testing.
- 5: Patients within a family with an negative/unknown TP53 mutation.

SUMMARY:
Background:

- Li-Fraumeni syndrome (LFS) is a genetic condition that increases the risk for some types of cancer. LFS may lead to cancer of the bone or connective tissue, breast, and brain. It may also increase the risk for certain types of leukemia and other cancers. The only known cause of LFS is a change (called a mutation ) in a gene known as TP53. However, not all people with LFS have a TP53 mutation. Researchers want to study other possible genetic causes of LFS, and factors that may increase or decrease cancer risk in people with the syndrome.

Objectives:

* To learn more about the types of cancers that occur in individuals with LFS.
* To study the role of the TP53 gene in the development of cancer.
* To look for other possible genes that cause LFS
* To study the effect of LFS diagnosis on families.
* To determine if environmental factors or other genes can change a person s cancer risk associated with LFS.

Eligibility:

* Individuals with a family or personal medical history of cancers consistent with LFS.
* Individuals with a family or personal medical history of cancers that does not meet the diagnosis of LFS, but the history is suggestive for LFS (meets the diagnosis for the so-called Li-Fraumeni like syndrome)
* Individuals with certain rare cancers
* Individuals with a family or personal history of a TP53 gene mutation, with or without related cancer(s).

Design:

* Participants will fill out a medical history questionnaire and a family history questionnaire.
* Blood samples will be collected for DNA and for storage. Cheek cell samples may be collected if blood cannot be obtained for DNA. Participants can choose to have or not have cancer screening with blood tests, imaging studies, and other exams.
* Participants will complete questionnaires about their worries about cancer, stress levels, and coping strategies. Diet and physical activity questionnaires will also be given. Other psychological tests may be given as needed.
* Participants will be monitored for several years, with regular followup visits to the National Institutes of Health, if indicated. Any changes in health or cancer status will be recorded.

DETAILED DESCRIPTION:
Study Description:

This is a natural history study involving questionnaires, clinical and research evaluations, clinical and research laboratory tests, review of

medical records, and cancer surveillance. This is a prospective long-term study of individuals at high risk of cancer due to Li-Fraumeni Syndrome (LFS) or Li-Fraumeni-Like Syndrome (LFL), using a cohort approach. Enrollees are invited to participate in all aspects of the study but can choose to opt out of specific part(s).

Objectives:

Primary Objectives:

* To ascertain/enroll individuals and families with Li-Fraumeni Syndrome (LFS) and Li-Fraumeni-Like Syndrome (LFL)
* To evaluation and define the clinical spectrum and natural history of disease in LFS and LFL
* To quantify cumulative cancer risk in individuals with LFS or LFL
* To develop a cancer screening program for individuals with LFS or LFL
* To investigate the mechanisms of tumorigenesis in LFS-related tumors (e.g., cell proliferation, growth regulation, apoptosis)
* To identify genetic determinants, environmental factors, and gene-environment interactions that potentially modify cancer risk in

these high-risk individuals

* To evaluate the psychological, behavioral, and social functioning effects of LFS on affected individuals and their family members
* To explore the plausibility of lifestyle interventions as potential strategies for cancer risk reduction
* To create an annotated biospecimen repository of LFS-related for translational, etiologic, and outcomes research

Secondary Objectives:

-To evaluate specific tumor characteristics, including histologies (e.g., leukemia types, brain tumor types, etc.) of cancers

diagnosed in individuals with LFS or LFL.

-To evaluate the potential effect of therapeutic radiation and radiation exposure from diagnostic/screening imaging studies on

cancer risk.

* To provide education, cancer risk assessment, and risk management recommendations for study participants.
* To collect clinical data related to the treatment of LFS-related cancers, so that outcome and survival may be evaluated.

Endpoints: Primary Endpoint:

-Occurrence of cancer in individuals and families with LFS or LFL

ELIGIBILITY:
* INCLUSION CRITERIA:
* On referral, persons of all ages will be considered for inclusion in the study

because of either:

* A family or personal medical history of neoplasia consistent with the diagnosis of LFS or LFL; or,
* A personal history of a germline TP53 mutation; or,
* A first- or second- degree relative of a TP53 mutation carrier, regardless of mutation status; or,
* A personal history of three or more LFS-related primary cancers; or,
* A personal history of adrenal cortical carcinoma or choroid plexus carcinoma at any age, regardless of family history

Personal and family medical history must be verified through questionnaires, interviews, review

of medical records and/or review of pathology slides.

There are 72 families who have previously enrolled in the pilot study under protocol 78-C-0039.

As the eligibility criteria remain the same, these families will be eligible for this protocol and will be invited to sign the new consent.

-Ability of subject or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document.

For both the Field and Clinical Center Cohort, the PI will ensure that study investigators will

identify an appropriate LAR consistent with requirements of Policy 403 and will obtain consent

from the LAR as outlined in the consent process before initiating research interventions.

-Pregnant women

In order to study the lifetime rates of cancer development in all individuals with Li-Fraumeni

syndrome, we will need to evaluate what effect pregnancy may have on rate of cancer

development both in affected individuals and unaffected family controls. Additionally, some

cancers are known to have an increased risk of development in the context of pregnancy and

lactation. Exclusion of pregnant women would preclude understanding of these cancer risks for

an important subset of the population.

Pregnant women are eligible for enrollment on the data collection component of this study.

Pregnant women will be included in this study as several endpoints may be assessed during

pregnancy; counseling, education, and other minimal risk procedures (i.e. blood draw) may be

done. We will postpone full clinical evaluations at the Clinical Center of pregnant women until

the subject has recovered post-partum.

All screening studies, for women who are pregnant, or breastfeeding will be deferred while the

woman is pregnant or breastfeeding. Pregnancy testing will be performed for females of childbearing age prior to imaging studies, and the test results must be negative prior to the scan..

The risk to the fetus and pregnant woman would be no greater than minimal for procedures that

are performed.

EXCLUSION CRITERIA:

* Referred individuals and families whose reported diagnoses cannot be verified
* Medical or psychiatric disorder which, in the opinion of the Principal Investigator, would preclude the ability to participate in clinical research
* Women who are pregnant will not be eligible for the cancer screening protocol until they recover post-partum. Women participating in the cancer screening protocol will discontinue this component if they become pregnant while on study. Once they recover post-partum, they can continue the cancer screening protocol.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Eligibility for the LFS study population: - A family or personal medical history of cancers consistent with the diagnosis of LFS or LFL; or, - A personal history of a germline TP53 mutation; or, - A first- or second- degree relative of a TP53 mutation carrier, regardless of mutation status; or, - A personal history of three or more LFS-related primary cancers; or, - A personal history of adrenal cortical carcinoma or choroid plexus carcinoma at any age
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2012-01-17 (Actual)

PRIMARY OUTCOMES:
Prevalence | ongoing
  Learn more about the types of cancers that occur in individuals with LFS and the age at which these cancers are usually found
Multiple measures | ongoing
  Explore ways to lower cancer risk
Multiple measures | ongoing
  Explore the typical features of the cancers diagnosed in individuals with LFS
Multiple measures | ongoing
  Explore the psychological and social functioning issues faced by LFS families
Multiple measures | ongoing
  Explore the best ways to look for cancers early in individuals with LFS
Multiple measures | ongoing
  Determine if there is any connection between specific mutations in the TP53 gene and the risk of certain type of cancers
Multiple measures | ongoing
  Determine if there are any environmental factors or other genes that can change a person's cancer risk associated with LFS
Multiple measures | ongoing
  Determine how often a change (mutation) in the TP53 gene is found in families in which LFS is suspected

CONTACTS AND LOCATIONS:
Overall Officials: Payal P Khincha, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - National Cancer Institute - Shady Grove, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland

REFERENCES:
- [Background] Mai PL, Malkin D, Garber JE, Schiffman JD, Weitzel JN, Strong LC, Wyss O, Locke L, Means V, Achatz MI, Hainaut P, Frebourg T, Evans DG, Bleiker E, Patenaude A, Schneider K, Wilfond B, Peters JA, Hwang PM, Ford J, Tabori U, Ognjanovic S, Dennis PA, Wentzensen IM, Greene MH, Fraumeni JF Jr, Savage SA. Li-Fraumeni syndrome: report of a clinical research workshop and creation of a research consortium. Cancer Genet. 2012 Oct;205(10):479-87. doi: 10.1016/j.cancergen.2012.06.008. Epub 2012 Aug 29. PMID 22939227
- [Background] Villani A, Tabori U, Schiffman J, Shlien A, Beyene J, Druker H, Novokmet A, Finlay J, Malkin D. Biochemical and imaging surveillance in germline TP53 mutation carriers with Li-Fraumeni syndrome: a prospective observational study. Lancet Oncol. 2011 Jun;12(6):559-67. doi: 10.1016/S1470-2045(11)70119-X. Epub 2011 May 19. PMID 21601526
- [Background] Malkin D. Li-fraumeni syndrome. Genes Cancer. 2011 Apr;2(4):475-84. doi: 10.1177/1947601911413466. PMID 21779515
- [Derived] Rising CJ, Huelsnitz CO, Shepherd RF, Klein WMP, Sleight AG, Wilsnack C, Boyd P, Feldman AE, Khincha PP, Werner-Lin A. Diet and physical activity behaviors: how are they related to illness perceptions, coping, and health-related quality of life in young people with hereditary cancer syndromes? J Behav Med. 2024 Aug;47(4):707-720. doi: 10.1007/s10865-024-00489-z. Epub 2024 Apr 20. PMID 38642305
- [Derived] Rising CJ, Wilsnack C, Boyd P, Sleight AG, Hutson SP, Khincha PP, Werner-Lin A. Family communication challenges of adolescents and young adults with Li-Fraumeni syndrome: Implications for psychosocial care. Patient Educ Couns. 2022 Nov;105(11):3259-3266. doi: 10.1016/j.pec.2022.07.012. Epub 2022 Jul 20. PMID 35918231
- [Derived] Werner-Lin A, Forbes Shepherd R, Young JL, Wilsnack C, Merrill SL, Greene MH, Khincha PP. Embodied risk for families with Li-Fraumeni syndrome: Like electricity through my body. Soc Sci Med. 2022 May;301:114905. doi: 10.1016/j.socscimed.2022.114905. Epub 2022 Mar 17. PMID 35367908
- [Derived] de Andrade KC, Khincha PP, Hatton JN, Frone MN, Wegman-Ostrosky T, Mai PL, Best AF, Savage SA. Cancer incidence, patterns, and genotype-phenotype associations in individuals with pathogenic or likely pathogenic germline TP53 variants: an observational cohort study. Lancet Oncol. 2021 Dec;22(12):1787-1798. doi: 10.1016/S1470-2045(21)00580-5. Epub 2021 Nov 12. PMID 34780712
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2011-C-0255.html